CLINICAL TRIAL: NCT05124821
Title: Evaluation of Performance Over Dwell Time and Safety of the Central-venous Catheters Certofix® Paed
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-2001
Record Dates: First submitted 2021-10-12; First posted 2021-11-18 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Central Venous Catheter
Keywords: Central Venous Catheter; Paediatrics; Post Marketing Clinical Follow-up; Seldinger Technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Certofix Paed: Paediatric patients in need for short-term (≤ 30 days) catheterisation of the superior vena cava using the Seldinger technique for infusion and volume therapy or parenteral nutrition, for administration of highly osmolar or very vein-irritating solutions/drugs, for continuous or intermittent monitoring of the central venous pressure, for blood sampling, or when peripheral venous puncture is not possible in state of shock, in patients with injured extremities or no detectable peripheral veins.
  Interventions: Device: Central venous catheter intended to be used for children during routine clinical practice

INTERVENTIONS:
Device: Central venous catheter intended to be used for children during routine clinical practice — Device will applied according to instruction for use (IFU) and respective indication during routine clinical practice.
  Other Names: Certofix® Paed

SUMMARY:
Central venous catheterisation is a medical technique that has become established over many decades and can be rated as State of the Art. However, there is only few clinical evidence for the use of Certofix® Paed and additional clinical data need to be collected to underline the long-term performance and safety in paediatric patients. An updated summary overview of Binninger and Roschke describes the potential incidence rates of the classically catheter-related complications, e.g. catheter malposition, catheter fracture, occlusion, thrombosis and catheter-related bloodstream infections (CRBSI) which may have an impact on overall morbidity, mortality and treatment costs. These catheter-related complications should be evaluated in this non-interventional study in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed assent from patients as well as written informed consent from legal representatives / parents (as applicable)
* Patient's first catheter placement during current hospital stay
* Placement of catheter according to IFU (Instruction for Use)

Exclusion Criteria:

* Contraindications according to IFU
* Patient has a documented or known allergy/sensitivity to a medical adhesive product such as transparent film, adhesive dressing, tapes or liquid skin protectants
* Inclusion in another interventional study in the field of central-venous catheters which could interfere with the routine clinical practice regarding the application and care of the product until removal

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients in need for short-term (≤ 30 days) catheterisation of the superior vena cava using the Seldinger technique for infusion and volume therapy or parenteral nutrition, for administration of highly osmolar or very vein-irritating solutions/drugs, for continuous or intermittent monitoring of the central venous pressure, for blood sampling, or when peripheral venous puncture is not possible in state of shock, in patients with injured extremities or no detectable peripheral veins.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Late complications | up to 30 days
  Incidence of thrombosis
Late complications | up to 30 days
  Incidence of occlusion
Late complications | up to 30 days
  Incidence of catheter insertion site infection
Late complications | up to 30 days
  Incidence of malpositioning of catheter due to dislodgement or migration

SECONDARY OUTCOMES:
Early complications of central venous catheter application | Up to 2 hours
Incidence of systemic infection | up to 30 days
Catheter handling details | up to 30 days
  Number of emergency applications of the catheter
Catheter handling details | up to 30 days
  Reason for insertion of catheter: infusion and volume therapy, parenteral nutrition, administration of highly osmolar solutions, administration of very vein-irritating solutions, continuous or intermittent monitoring of the central venous pressure, peripheral venous puncture was not successful or veins not detectable
Catheter handling details | up to 30 days
  Place of positioning of catheter
Catheter handling details | up to 30 days
  Ultrasound guided central venous catheter application
Catheter handling details | up to 30 days
  Control of catheter positioning: radiologic, ECG
Catheter handling details | up to 30 days
  Date of catheter insertion and removal
Catheter handling details | up to 30 days
  Time of catheter insertion and removal
Catheter handling details | up to 30 days
  Catheter fixation
Catheter handling details | up to 30 days
  Catheter Care
Catheter handling details | up to 30 days
  Observations on catheter quality
Concomitant medication | up to 30 days
  Use of antibiotics or other relevant medication
Adverse Device Effect (ADE) | up to 30 days
Device Deficiency (DD) | up to 30 days
  Device deficiency
Device Deficiency (DD) | up to 30 days
  Duration of device deficiency
Device Deficiency (DD) | up to 30 days
  Action taken
Serious Adverse Event (SAE) | up to 30 days
Serious Adverse Device Effect (SADE) | up to 30 days
Catheter variables | up to 30 days
  Number of lumen
Catheter variables | up to 30 days
  Size
Catheter variables | up to 30 days
  Length
Reason for removal of catheter | up to 30 days
  Regular end of infusion therapy or removal according to local standards
Reason for removal of catheter | up to 30 days
  Upcoming sings of infection on puncture site: skin reddening, swelling, pain, increased skin temperature, fever with unclear origin, other
Reason for removal of catheter | up to 30 days
  Early complication
Reason for removal of catheter | up to 30 days
  Late complication
Reason for removal of catheter | up to 30 days
  Technical problems with the catheter
Demographic data | Prior study start
  Age
Demographic data | Prior study start
  Sex
Demographic data | Prior study start
  Ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sasse, Dr. med., Study Chair — Hannover Medical School
Locations (3):
- Medizinische Hochschule Hannover, Klinik für Pädiatrische Kardiologie und Pädiatrische Intensivmedizin, Hanover, Germany
- Italy (2):
  - Istituto Giannina Gaslini, Anesthesia and Acute and Procedural Pain Therapy, Genova
  - Ospedale de Bambini Vittore Buzzi, Milan

IPD SHARING:
Plan to Share IPD: No